CLINICAL TRIAL: NCT01937143
Title: Immunizing Infants Against Pain: a Hospital-based Postnatal Parent Education Intervention About Infant Immunizations
Brief Title: A Hospital-based Postnatal Parent Education Intervention About Infant Immunizations
Acronym: IIAP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Toronto (Other)
Responsible Party: Principal Investigator, Anna Taddio, Professor, Leslie Dan Faculty of Pharmacy, University of Toronto
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 126007; 126007 (Other Grant/Funding Number: Canadian Institutes of Health Research)
Record Dates: First submitted 2013-08-26; First posted 2013-09-09 (Estimated); Last update posted 2016-09-21 (Estimated); Status verified 2016-09

CONDITIONS: Postpartum Women
Keywords: parent education; immunization; vaccination; infant; pain management
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Control (Placebo Comparator): General information about infant immunizations at birth of a newborn infant
  Interventions: Behavioral: Control
- Low intensity intervention (Active Comparator): Pamphlet with information about pain management during infant immunizations at birth of a newborn infant
  Interventions: Behavioral: Low intensity intervention
- High intensity intervention (Active Comparator): Pamphlet and video with information about pain management during infant immunizations at birth of a newborn infant
  Interventions: Behavioral: High intensity intervention

INTERVENTIONS:
Behavioral: Low intensity intervention — Pamphlet with information about pain management during infant immunizations at birth of a newborn infant
  Arms: Low intensity intervention
Behavioral: High intensity intervention — Pamphlet and video with information about pain management during immunizations at birth of a newborn infant
  Arms: High intensity intervention
Behavioral: Control — General information about infant immunizations at birth of a newborn infant
  Arms: Control

SUMMARY:
Immunization injections are the most common recurring painful medical procedure undertaken in childhood. Numerous evidence-based and feasible interventions are available to mitigate immunization pain, however, there is low uptake of these interventions in clinical practice, revealing a knowledge-to-care gap between what is known about pain and pain management. This is a 4-year single-centre, randomized, parallel 3-group add-on trial that will enrol 3420 mothers hospitalized following the birth of an infant at Mount Sinai Hospital (MSH) in Toronto. The trial will evaluate and compare the impact of two levels of intensity of maternal education about pain management during infant immunizations ('low': pamphlet vs. 'high': pamphlet + video) compared to placebo control after the birth of an infant on maternal behaviour during future infant immunizations at up to 6 months of age (use of analgesic interventions), maternal knowledge and attitudes about pain and pain management up to 6 months after birth.

ELIGIBILITY:
Inclusion Criteria:

* mothers rooming in with infants on postnatal ward

Exclusion Criteria:

* mothers with significant psychiatric conditions
* mothers unable to communicate in English
* mothers sharing room whereby another mother already participated

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3420 (Estimated)
Dates: Start 2013-10; Primary Completion 2017-08 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Analgesic utilization | Up to 6 months
  Parent self-reported use of any of the 3 most effective analgesic interventions (breastfeeding, sugar water, or topical anesthetics) at infant immunization; the specific time period for the outcome assessment is at either 2, 4 or 6 month infant immunization, based on a random allocation process.

SECONDARY OUTCOMES:
Knowledge | Up to 6 months
  Parent knowledge about effective analgesic interventions for mitigating pain at infant immunization; the specific time period for the outcome assessment is at either 2, 4 or 6 month infant immunization, based on a random allocation process.
Attitudes | Up to 6 months
  Parent self-reported attitudes about pain/pain management at infant immunization; the specific time period for the outcome assessment is at either 2, 4 or 6 month infant immunization, based on a random allocation process.
Specific analgesic utilization | Up to 6 months
  Parent self-reported utilization of specific analgesic interventions at infant immunization; the specific time period for the outcome assessment is at either 2, 4 or 6 month infant immunization, based on a random allocation process.
Immunization compliance | Up to 6 months
  Parent self-reported compliance with infant immunization schedule, confirmed with health care provider if possible.

OTHER OUTCOMES:
Attempted analgesic utilization | Up to 6 months
  Parent self-reported attempted (and failed) use of any of the 3 most effective analgesic interventions (breastfeeding, sugar water, or topical anesthetics) at infant immunization; the specific time period for the outcome assessment is at either 2, 4, or 6 month infant immunization, based on a random allocation process.

CONTACTS AND LOCATIONS:
Overall Officials: Anna Taddio, PhD, Principal Investigator — University of Toronto
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Taddio A, Shah V, Bucci L, MacDonald NE, Wong H, Stephens D. Effectiveness of a hospital-based postnatal parent education intervention about pain management during infant vaccination: a randomized controlled trial. CMAJ. 2018 Oct 22;190(42):E1245-E1252. doi: 10.1503/cmaj.180175. PMID 30348739